CLINICAL TRIAL: NCT03108105
Title: Multicenter Pilot Study to Describe the Performance of the AOS-C2001-B Device in Patients With Colostomy
Brief Title: Multicenter Study to Describe the Performance of the AOS-C2001-B Device in Patients With Colostomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BBraun Medical SAS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OPM-G-H-1604
Record Dates: First submitted 2017-04-05; First posted 2017-04-11 (Actual); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Colostomy Stoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AOS-C2001-B (Experimental): A new 2-piece appliance composed with 2 parts: a base plate and an ostomy collection special pouch (1 base plate for 2 or 3 days and 1 to 4 collection special pouch per day)
  Interventions: Device: AOS-C2001-B

INTERVENTIONS:
Device: AOS-C2001-B — A new 2-piece appliance composed with 2 parts: a base plate and an ostomy collection special pouch (1 base plate for 2 or 3 days and 1 to 4 collection special pouch per day)

SUMMARY:
The study evaluates the efficacy of a new 2-piece appliance in patients with colostomy.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 years old
* Patient having a colostomy with a diameter less than 30 mm for users of Ø 55 mm pouches or having a colostomy with a diameter less than 40 mm for users of Ø 65 mm pouches
* Patient having a colostomy for at least 1 month
* Patient using a flat ostomy appliance
* Patient having a stoma protusion smaller than or equal to 1.5 cm
* Patient capable to apply and remove the appliance himself or with the help of a caregiver (except health care professional)
* Patient having a mental capacity to participate to the study (i.e. to understand the study and to answer to the questions)
* Patient agreeing to test the new appliance during the evaluation phase (14±3 days)
* Patient covered by social security

Exclusion Criteria:

* Patient experiencing repeated leakages with the usual pouching system
* Patient currently suffering from peristomal skin complications (bleeding or red and broken skin at the time of inclusion)
* Patient receiving or having received, within the last month, chemotherapy, radiotherapy or corticotherapy
* Patient already participating in another clinical study or who have previously participated in this investigation
* Pregnant or breast-feeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-11-07 (Actual); Study Completion 2017-11-07 (Actual)

PRIMARY OUTCOMES:
Description of efficacy in terms of stool collection and leakage prevention | At least 1 time per day during 14±3 days
  After each change of the investigational product, the patient will describe on a 4-point scale the type of capsule cap cover removal
Description of efficacy in terms of stool collection and leakage prevention | At least 1 time per day during 14±3 days
  After each change of the investigational product, the patient will describe on a 4-point scale the level of leakage

CONTACTS AND LOCATIONS:
Locations (1):
- Elie CHOUILLARD, Poissy, France

IPD SHARING:
Plan to Share IPD: No